CLINICAL TRIAL: NCT01868854
Title: Risk Assessment of Peritoneal Dialysis Failure Based on Catheter Tip Location. Multicentric Study.
Brief Title: Risk Assessment of Peritoneal Dialysis Failure Based on Catheter Tip Location.
Acronym: TIP-DP
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Collaborators: JOSE CARRASCO ARTEAGA HOSPITAL FROM Ecuadorian Institute of Social Security (Unknown); Hospital de Especialidades de las Fuerzas Armadas HE 1 QUITO (Unknown)
Responsible Party: Principal Investigator, FRANKLIN MORA, MD, Instituto Nacional de Cardiologia Ignacio Chavez
Other Study IDs: Incich-2013-Dp-0012
Record Dates: First submitted 2013-04-22; First posted 2013-06-05 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-05

CONDITIONS: Renal Failure
Keywords: Tip catheter; Peritoneal Dialysis; Risk Factot; Mecanical Function
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Radiographic Plane 1: the tip of peritoneal dialysis catheter is located at the bottom of the pelvis, below a line connecting the head of the femur
- Radiographic Plane 2: the tip of the peritoneal dialysis catheter is located above the plane 1 and below a line connecting the two iliac spines
- Radiographic plane 3: The location of the catheter tip is on the line connecting iliac spines and below a line connecting the iliac crests
- Radiographic plane 4: The location of the catheter tip is on the line connecting the iliac crests

SUMMARY:
The location of the catheter tip in radiographic planes 1 and 2, is a protection factor for the mechanical performance of peritoneal Dialysis. Instead radiographic planes 3 and 4 are risk factors.

DETAILED DESCRIPTION:
Radiolucency of the peritoneal dialysis catheter, allow to classify the location of the tip into 4 radiographic planes. Plane 1: below the zone of a line on the head of the femur. Plane 2: is the area above the plane 1 and below a line connecting the two iliac spines. Plane 3: is the area that is above the plane 2 and below a line connecting the upper edge of the two iliac crests. Plane 4: is the area located above the plane 3.

ELIGIBILITY:
Inclusion Criteria:

* patients with functional class K-Digo 5d, initiating peritoneal dialysis program, with recent positioning of less than 2 weeks of dialysis catheter placement

Exclusion Criteria:

* patients with agenesis of pelvic bones that prevent divisions radiographic

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic renal failure 5d: who are initiating peritoneal dialysis in any form
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-12 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
MECHANICAL OPERATION OF PERITONEAL DIALYSIS CATHETER | TWELVE HOURS AFTER CATHETER PLACEMENT
  MEASURE THE TIME THAT RETURNING IN 1 LITER OF SOLUTION AFTER INFUSION PERITONEAL. TAKE IT AS FLUID RETURN FAILURE WHEN A DELAY SAME OR GREATER THAN 20 MINUTES.

SECONDARY OUTCOMES:
LOCATION OF THE TIP OF PERITONEAL DIALYSIS CATHETER THROUGH STANDING ABDOMINAL RADIOGRAPHY | 12 HOURS AFTER CATHETER PLACEMENT, AND THE PATIENT WILL BE OBSERVED BY 1 WEEK
  RADIOGRAPIC PLANS ARE CLASSIFIED IN 4 LEVEL: 1) BELOW THE "HEADS OF THE FEMUR", 2) BELOW " ILIAC SPINES", 3) BELOW THE "ILIAC CREST", 4) ABOVE "THE ILIAC CREST".

OTHER OUTCOMES:
DESCRIPTIVE VARIABLES | PARTCIPANTS WILL BE FOLLOWED FOR THE DURATION OF HOSPITAL STAY, AND EXPECTED AVERAGE OF 2 WEEKS
  WEIGHT, SIZE, SEX, DIAGNOSIS, KT / V, AMONG OTHER

CONTACTS AND LOCATIONS:
Overall Officials: Franklin Mora, MD, Study Director — "José Carrasco Arteaga" Hospital, Cuenca-Ecuador.; Jorge Huertas, MD, Principal Investigator — Hospital de Especialidades de las Fuerzas Armadas. Quito (Ecuador); Magdalena Madero, MSC, Principal Investigator — "INSTITUTO NACIONAL IGNACIO CHAVEZ" México D.F.; Oscar Hernández, MD, Principal Investigator — "Instituto Nacional de Cardiología Ignacio Chávez".; Juan F Herrera, MD, Principal Investigator — Centro Médico ABC, Methodist International, Mexico D.F.; Alfonso Mariscal, MSC, Principal Investigator — Hospital Civil, Morelia Michoacán, México; Guadalupe De LA Cruz, RN, Principal Investigator — Hospital José Carrasco Arteaga, Cuenca-Ecuador

REFERENCES:
- [Background] De La Cruz G, Mora-Bravo F. Novel Classification to Monitor the Location of Peritoneal Dialysis Catheters. Blood Purif 35: 160-1, 2013.